CLINICAL TRIAL: NCT03014895
Title: A Randomized, Double-blind, Placebo-controlled, Single Intravenous Ascending Dose Study of E3112 in Japanese Healthy Adult Male Subjects
Brief Title: A Single Intravenous Dose Study of E3112 in Japanese Healthy Adult Male Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: EA Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: E3112/CP1
Record Dates: First submitted 2017-01-06; First posted 2017-01-09 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-06

CONDITIONS: Healthy Male Volunteers
Keywords: E3112; Pharmacokinetics; Japanese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort 1: Placebo (Placebo Comparator): Intravenous placebo infusion
  Interventions: Drug: Placebo
- Cohort 1: E3112 (Experimental): Intravenous E3112 infusion
  Interventions: Drug: E3112
- Cohort 2: Placebo (Placebo Comparator): Intravenous placebo infusion
  Interventions: Drug: Placebo
- Cohort 2: E3112 (Experimental): Intravenous E3112 infusion
  Interventions: Drug: E3112
- Cohort 3: Placebo (Placebo Comparator): Intravenous placebo infusion
  Interventions: Drug: Placebo
- Cohort 3: E3112 (Experimental): Intravenous E3112 infusion
  Interventions: Drug: E3112
- Cohort 4: Placebo (Placebo Comparator): Intravenous placebo infusion
  Interventions: Drug: Placebo
- Cohort 4: E3112 (Experimental): Intravenous E3112 infusion
  Interventions: Drug: E3112
- Cohort 5: Placebo (Placebo Comparator): Intravenous placebo infusion
  Interventions: Drug: Placebo
- Cohort 5: E3112 (Experimental): Intravenous E3112 infusion
  Interventions: Drug: E3112

INTERVENTIONS:
Drug: Placebo — Intravenous infusion
  Arms: Cohort 1: Placebo; Cohort 2: Placebo; Cohort 3: Placebo; Cohort 4: Placebo; Cohort 5: Placebo
Drug: E3112 — Intravenous infusion
  Arms: Cohort 1: E3112; Cohort 2: E3112; Cohort 3: E3112; Cohort 4: E3112; Cohort 5: E3112

SUMMARY:
The study (E3112/CP1) is a single-center, randomized, double-blind, placebo-controlled, single intravenous ascending dose study conducted in Japanese healthy adult males to evaluate the pharmacokinetics (PK), safety, and immunogenicity of E3112 following a single intravenous dose of E3112.

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion Criteria:

* Non-smoking, Japanese, male participants, ≥20 and <45 years old at the time of obtaining informed consent
* Have a Body Mass Index (BMI) ≥18.5 and <25.0 kilograms per meters squared (kg/m^2) at Screening
* Able to provide written informed consent of their free will
* Males who were given a full explanation of all the requirements of the protocol, and are willing and able to comply with them

Exclusion Criteria:

Main Exclusion Criteria:

* Male and his partner who do not agree to use a highly effective method of contraception throughout the entire study period, if he has reproductive capacity
* Male who had or has any malignant tumor, lymphoma, leukaemia, or lymphoproliferative disorders. Clinically significant illness that required medical treatment within 8 weeks or a clinically significant infection within 4 weeks prior to dosing.
* Evidence of disease that may influence the outcome of the study within 4 weeks prior to dosing
* Any history of surgical treatment that may affect pharmacokinetic (PK) profiles of study drug at Screening
* Any suspected clinically abnormal symptom or organ impairment that require medical treatment at Screening or Baseline
* Receipt of vaccination within 4 weeks prior to dosing
* History of drug or alcohol dependency or abuse prior to Screening
* Intake of caffeinated beverages or food within 72 hours prior to dosing
* Use of prescription drugs within 4 weeks prior to dosing
* Intake of over-the-counter (OTC) medications within 2 weeks prior to dosing
* Male who is currently being enrolled in another clinical study or used any investigational drug or device in another clinical study within 16 weeks prior to dosing
* Male who underwent a blood transfusion within 12 weeks prior to dosing, who donate 400 milliliters (mL) or more of whole blood within 12 weeks prior to dosing, who donate 200 mL or more of whole blood within 4 weeks prior to dosing, or who made a component donation within 2 weeks prior to dosing

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-11-22 (Actual)

PRIMARY OUTCOMES:
Peak concentration (Cmax) of E3112 | Days 1 to 4, 8, 14, and 28
  Cmax is the maximum observed concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administered.
Time to peak concentration (Tmax) of E3112 | Days 1 to 4, 8, 14, and 28
  Tmax is the time from dosing to reach the maximum observed concentration a drug achieves in a specified compartment or test area of the body after the drug has been administered.
Area under the curve (AUC) | Days 1 to 4, 8, 14, and 28
  AUC is the area under the curve in a plot of concentration of drug in blood plasma against time. AUC represents the total drug exposure over a defined period of time.
Half-life of elimination (t1/2) of E3112 | Days 1 to 4, 8, 14, and 28
  t1/2 is the time required for the concentration of the drug to reach half of its original value.
Clearance of E3112 | Days 1 to 4, 8, 14, and 28
  Clearance is defined as the rate of drug elimination divided by the plasma concentration of the drug.
Volume of distribution (Vd) of E3112 | Days 1 to 4, 8, 14, and 28
  Vd is the theoretical volume that would be necessary to contain the total amount of an administered drug at the same concentration that it is observed in the blood plasma.

SECONDARY OUTCOMES:
Number of participants with any serious adverse event and any non-serious adverse event | Days 1 to 28
  An adverse event is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A serious adverse event is defined as any adverse event occurring at any dose that results in any of the following outcomes: results in death; is life threatening; results in inpatient hospitalization or prolongation of existing hospitalization; results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life function; results in a congenital anomaly/birth defect; or can be defined as any other important medical event.
Number of participants with an abnormal, clinically significant hematology parameter value | Days 1 to 28
  Clinical significance will be determined by the investigator.
Number of participants with an abnormal, clinically significant blood chemistry parameter value | Days 1 to 28
  Clinical significance will be determined by the investigator.
Number of participants with an abnormal, clinically significant urine value | Days 1 to 28
  Clinical significance will be determined by the investigator.
Number of participants with an abnormal, clinically significant vital sign measurement | Baseline; Days 1 to 28
  Clinical significance will be determined by the investigator.
Number of participants with an abnormal, clinically significant electrocardiogram (ECG) measurement | Baseline; Days 1 to 28
  Clinical significance will be determined by the investigator.
Number of participants with an abnormal, clinically significant physical examination measurement | Baseline; Days 1 to 28
  Clinical significance will be determined by the investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- EA Pharma Trial Site, Toshima City, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No